CLINICAL TRIAL: NCT03662776
Title: Effect of Treatment Modality on Psychosocial Functioning of Survivors of Unilateral Retinoblastoma
Status: Enrolling by invitation | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 18-397
Record Dates: First submitted 2018-09-04; First posted 2018-09-07 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Survivors of Unilateral Retinoblastoma
Keywords: Quality of Life; physical health; emotional health; 18-397
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- retinoblastoma survivors treated with enucleation: MSK will contact all families of 1-year survivors of unilateral retinoblastoma treated with enucleation or intra-arterial chemotherapy at MSK and TCH between 2006 or later for completion of validated questionnaires integrating the BASC-3 and PROMIS surveys. The survey may be administered in-person during clinic or by mail, based upon participant preference.
  Interventions: Behavioral: BASC-3 survey; Behavioral: PROMIS survey
- retinoblastoma survivors treated with intra-arteria chemo: MSK will contact all families of 1-year survivors of unilateral retinoblastoma treated with enucleation or intra-arterial chemotherapy at MSK and TCH between 2006 or later for completion of validated questionnaires integrating the BASC-3 and PROMIS surveys. The survey may be administered in-person during clinic or by mail, based upon participant preference.
  Interventions: Behavioral: BASC-3 survey; Behavioral: PROMIS survey

INTERVENTIONS:
Behavioral: BASC-3 survey — A comprehensive questionnaire, incorporating the BASC-3 and PROMIS measures, will be administered to parents of participants ages 8-17. The BASC-3 and PROMIS scales each have a parent and child version; these scales will be used to measure the secondary objective of parent and patient concordance rates for all participants ages 8 and older.
Behavioral: PROMIS survey — A comprehensive questionnaire, incorporating the BASC-3 and PROMIS measures, will be administered to parents of participants ages 8-17. The BASC-3 and PROMIS scales each have a parent and child version; these scales will be used to measure the secondary objective of parent and patient concordance rates for all participants ages 8 and older.

SUMMARY:
The purpose of this study is to find out about the quality of life and health in patients who had retinoblastoma in one eye (unilateral retinoblastoma), who either received treatment with chemotherapy injected directly into an artery leading to the eye (intra-arterial chemotherapy) or removal of the eye (enucleation). By quality of life, the investigators mean how the participants are feeling about being satisfied with things in their life, including, physical health, emotional health, and their ability to carry out daily activities. The investigators want to see if either treatment option would affect quality of life differently. The investigators hope that this information will help us provide better care to future children with retinoblastoma and better follow-up care for survivors of retinoblastoma.

ELIGIBILITY:
Inclusion Criteria:

* Ability to speak and understand English or Spanish
* Diagnosis of unilateral retinoblastoma at any age, confirmed by the enrolling institution
* Treatment of retinoblastoma between 2006 or later
* Patients must between the age of 8-17 years old
* At least 1 year since completion of all cancer-directed therapy
* Treatment with enucleation of the affected eye or intra-arterial chemotherapy

Parent of patient:

* Ability to speak and understand English or Spanish
* Ability to confirm that he or she is the parent of a child treated for unilateral retinoblastoma who meets the eligibility criteria listed above
* Ability to provide informed consent

Exclusion Criteria:

* Patients, or parents of patients, treated with both enucleation and intra-arterial chemotherapy are not eligible

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Eligible survivors of unilateral retinoblastoma will be identified via the MSK and TCH databases and offered participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-08-31 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
social-emotional health | 2 years
  as measured by Behavior Assessment System for Children, 3rd edition, (BASC™-3;as measured by the BASC-3) Surveys have been normed on a representative sample that closely matches United States census population characteristics; T scores and percentiles in relation to general norms are calculated for each scale. The BASC-3 uses a T score metric where 50 is the mean for the population norm and the standard deviation is 10.
behavioral health | 2 year
  as measured by Behavior Assessment System for Children, 3rd edition, (BASC™-3; The following four T Scores will be analyzed for these BASC-3 summary scores (1) Externalizing Problems, (2) Internalizing Problems, (3) Behavior Symptoms Index and (4) Adaptive Skills. The "at-risk" category applies to any individual who scores 2 SD above the mean of 50, while "clinically significant" risk refers to those who score 3 SD above the mean. Additional scores are also provided which may be used to identify risk for more specific behavioral or emotional areas of concern.
compare HRQoL | 2 years
  as measured by the Patient Reported Outcomes Measurement Information System (PROMIS®) PROMIS measures use a T-score metric where 50 is the mean for the reference population and 10 is the standard deviation of that population. Higher scores correspond to a higher degree of symptom burden (for those items measuring symptoms) or a higher level of functioning (for physical functioning items)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Cimini, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Texas Children's Hospital (Data Collection), Houston, Texas

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm